CLINICAL TRIAL: NCT01534715
Title: A Phase I, Multi-center, Open-label Study of IMGN529 Administered Intravenously in Adult Patients With Relapsed or Refractory Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: IMGN529 in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma and Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMGN0301
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2016-08

CONDITIONS: Lymphoma, Non-Hodgkin; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — naratuximab emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMGN529 (Experimental): Dose escalation study, dosing done every 3 weeks.
  Interventions: Drug: IMGN529

INTERVENTIONS:
Drug: IMGN529

SUMMARY:
The purpose of this study is to test the safety and tolerability of IMGN529 in patients with relapsed or refractory non-Hodgkin's lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory NHL including tumor types: Follicular lymphoma (FL), marginal zone lymphoma (MZL)/mucosa-associated lymphoid tissue (MALT), diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma (MCL), chronic lymphocytic leukemia (CLL).
* Adequate organ function
* ECOG ≤ 2
* Recovered or stabilized from prior treatments.

Exclusion Criteria:

* Allogeneic stem cell transplantation
* Pregnant or lactating females
* Known central nervous system, meningeal or epidural disease including brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities | During study

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - CTRC at UTHSCSA, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Oncology Institute of Southern Switzerland, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No